CLINICAL TRIAL: NCT04773925
Title: The Impact of Integrative Medicine on Patient-Reported Outcomes in Management of Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aakriti R. Carrubba, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-000221
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Chronic Female Pelvic Pain Syndrome (Disorder)

STUDY DESIGN:
Intervention Model Description: Women with chronic pelvic pain will be recruited during outpatient visits to Mayo Clinic Florida. Baseline patient-reported outcomes will be obtained using the PROMIS-CAT questionnaire. Questionnaires will be assigned in the electronic medical record. All subjects will receive standard care for their chronic pelvic pain, including a consultation with a gynecologist. Patients will then be referred for three 60-minute mindfulness counseling sessions conducted via telemedicine with a certified Mind-Body Counselor who has a degree in Social Work in the department of Integrative Medicine. The initial consultation will consist of a 60-minute individual session. The subsequent sessions will be group visits (anticipate 5 subjects per group) lasting 60 minutes. PROMIS-CAT questionnaires will be repeated at 3 months and 6 months, and a satisfaction survey will be distributed at the completion of the program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness group (Experimental): As this is a pilot feasibility trial, there is only one arm. All subjects will receive the mindfulness intervention if they consent to participate in the study.
  Interventions: Behavioral: Mindfulness counseling

INTERVENTIONS:
Behavioral: Mindfulness counseling — Subjects three 60-minute mindfulness counseling sessions with a certified Mind-Body Counselor who has a degree in Social Work in the department of Integrative Medicine. The mindfulness sessions will be conducted entirely via telemedicine. The initial consultation will consist of a 60-minute individual session. The next session will be a group visit (plan for 5 subjects per group) lasting 60 minutes, which will be scheduled for 2 weeks after the initial session. The third session will be another 60-minute group session, which will be scheduled for 6 weeks after the initial session.

SUMMARY:
The purpose of this research is to determine if mind and body counseling and training improves quality of life in women undergoing treatment for chronic pelvic pain.

DETAILED DESCRIPTION:
Patients with chronic illnesses are expected to self-manage much of their treatment. Barriers include limited time during appointments, consultations with multiple different providers, technical communication style, health literacy issues, and a sense of feeling overwhelmed. Patients with chronic pain syndromes experience symptoms which can negatively impact their quality of life by interfering with ability to sleep, work, and function in their social roles. One proposed mechanism in chronic pain management is mindfulness. Mindfulness is the intentional and non-judgmental conscious awareness of the present moment, or "paying attention on purpose" with the goal of physical and psychological health improvement. Participants are taught autonomy, increasing self-regulation, and focusing awareness on a particular goal or activity.

The investigators hypothesize that a mind-body counselor will improve patient engagement and promote adherence to pain coping treatments. If the initial findings from this project support the use of Integrative Medicine services in women with chronic pelvic pain, the investigators hope to expand this study to a larger, randomized controlled trial that is adequately powered to determine significant difference among participants in the control and study groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic pelvic pain.
* Must speak English.
* Must be ages 18 through 89.
* Must be willing and able to provide informed consent for participation.
* Must have access to the Patient Online Services portal to complete the questionnaires.

Exclusion Criteria:

- Diagnoses of primarily non-gynecologic pain, acute pelvic pain, and active abdominal or pelvic malignancy.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with improved quality of life scores on PROMIS-CAT questionnaires after treatment of chronic pelvic pain and enrollment in a mind-body training program | 6 months
  This outcome measure will demonstrate whether the proposed intervention showed improvement in symptomatology of subjects with chronic pain.

SECONDARY OUTCOMES:
Number of participants who were able to attend all mind-body training sessions | 6 months
  This outcome measure will be used to determine adherence and attendance to the Integrative Medicine services.
Time from enrollment in the study until completion of all mind-body sessions | 6 months
  This outcome measure will determine feasibility of scheduling patients with Integrative Medicine services and determine waiting list times for this service.

CONTACTS AND LOCATIONS:
Overall Officials: Aakriti R Carrubba, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- [Background] Alders I, Smits C, Brand P, van Dulmen S. Does patient coaching make a difference in patient-physician communication during specialist consultations? A systematic review. Patient Educ Couns. 2017 May;100(5):882-896. doi: 10.1016/j.pec.2016.12.029. Epub 2016 Dec 29. PMID 28089309
- [Background] Lachance CC, McCormack S. Mindfulness Training and Yoga for the Management of Chronic Non-malignant Pain: A Review of Clinical Effectiveness and Cost-effectiveness [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2019 Sep 20. Available from http://www.ncbi.nlm.nih.gov/books/NBK549581/ PMID 31725209
- [Background] Crisp CD, Hastings-Tolsma M, Jonscher KR. Mindfulness-Based Stress Reduction for Military Women With Chronic Pelvic Pain: A Feasibility Study. Mil Med. 2016 Sep;181(9):982-9. doi: 10.7205/MILMED-D-15-00354. PMID 27612341
- [Background] Ball EF, Nur Shafina Muhammad Sharizan E, Franklin G, Rogozinska E. Does mindfulness meditation improve chronic pain? A systematic review. Curr Opin Obstet Gynecol. 2017 Dec;29(6):359-366. doi: 10.1097/GCO.0000000000000417. PMID 28961631
- [Background] Jaderek I, Lew-Starowicz M. A Systematic Review on Mindfulness Meditation-Based Interventions for Sexual Dysfunctions. J Sex Med. 2019 Oct;16(10):1581-1596. doi: 10.1016/j.jsxm.2019.07.019. PMID 31570137
- [Background] Brotto LA, Basson R, Luria M. A mindfulness-based group psychoeducational intervention targeting sexual arousal disorder in women. J Sex Med. 2008 Jul;5(7):1646-59. doi: 10.1111/j.1743-6109.2008.00850.x. PMID 18507718
- [Background] Ball E, Newton S, Kahan BC, Forbes G, Wright N, Cantalapiedra Calvete C, Gibson HAL, Rogozinska E, Rivas C, Taylor SJC, Birch J, Dodds J. Smartphone App Using Mindfulness Meditation for Women With Chronic Pelvic Pain (MEMPHIS): Protocol for a Randomized Feasibility Trial. JMIR Res Protoc. 2018 Jan 15;7(1):e8. doi: 10.2196/resprot.7720. PMID 29335232
- [Background] Forbes G, Newton S, Cantalapiedra Calvete C, Birch J, Dodds J, Steed L, Rivas C, Khan K, Rohricht F, Taylor S, Kahan BC, Ball E. MEMPHIS: a smartphone app using psychological approaches for women with chronic pelvic pain presenting to gynaecology clinics: a randomised feasibility trial. BMJ Open. 2020 Mar 12;10(3):e030164. doi: 10.1136/bmjopen-2019-030164. PMID 32165549
- [Background] Brotto LA, Bergeron S, Zdaniuk B, Driscoll M, Grabovac A, Sadownik LA, Smith KB, Basson R. A Comparison of Mindfulness-Based Cognitive Therapy Vs Cognitive Behavioral Therapy for the Treatment of Provoked Vestibulodynia in a Hospital Clinic Setting. J Sex Med. 2019 Jun;16(6):909-923. doi: 10.1016/j.jsxm.2019.04.002. Epub 2019 May 15. PMID 31103481
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials